CLINICAL TRIAL: NCT06441435
Title: To Investigate the Protective Effect of AC 134 in Chronic Kidney Diseases.
Brief Title: The Effect of AC-134 in Chronic Kidney Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: All Clean Health Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SF23520C
Record Dates: First submitted 2024-05-21; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Nephrology
Keywords: Chronic Kidney Diseases; Activated charcoal
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anthrax | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Low-protein diet strategies combined with AC-134 capsules
  Interventions: Dietary Supplement: Low protein diet with AC-134
- Control group (Active Comparator): Low-protein diet strategies
  Interventions: Other: Standard treatment

INTERVENTIONS:
Dietary Supplement: Low protein diet with AC-134 — Low protein diet combined with AC-134 Dosage: 2 capsules,three times/day
  Arms: Intervention group
Other: Standard treatment — Low protein diet
  Arms: Control group

SUMMARY:
The objective is to explore the effects of adding AC-134 on renal function, proteinuria, uremic toxins, and metabolism-related markers in chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) management primarily focuses on addressing associated complications such as hypertension, diabetes mellitus, cardiovascular disease, and proteinuria. In addition to standard therapies, reducing the accumulation of toxins, particularly gut-derived uremic toxins like indoxyl sulfate (IS) and p-cresol sulfate (PCS), may help alleviate uremia symptoms. This study assesses the impact of oral AC-134 capsules containing activated charcoal adsorbent on CKD patients. The assessment will include evaluating changes in renal function, proteinuria, uremic toxins, and metabolism-related markers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-90 years.
* Diagnosed with stage 3-5 chronic kidney disease, excluding dialysis patients.
* Signed informed consent is required before enrollment.

Exclusion Criteria:

* Use of other brand-activated charcoal supplements during the study period.
* Pregnant or lactating women.
* Patients who have undergone kidney transplantation.
* Obstructive nephropathy within the past month.
* Acute kidney injury within the past three months.
* Gastrointestinal bleeding or severe constipation within the past three months.
* Patients with active malignancy within the past two years.
* Severe cardiovascular diseases such as congestive heart failure New York class III-IV or cerebrovascular disease
* Severe liver disease, such as liver cirrhosis with ascites.
* Active infectious disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-24 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) measurement | Baseline to 3 months
  The eGFR level is a maker for kidney function
Blood Urea Nitrogen (BUN) levels | Baseline to 3 months
  Blood Urea Nitrogen
Uremic toxins assay | Baseline to 3 months
  The concentration of p-cresol sulfate level, indoxyl sulfates level, and acrolein in the subjects' blood samples

SECONDARY OUTCOMES:
Liver function | Baseline to 3 months
  The concentration of ALT, AST, total bilirubin and direct bilirubin in the subjects' blood samples
Inflammation makers | Baseline to 3 months
  The concentration of inflammation makers in the subjects' blood samples
Nutrition status | Baseline to 3 months
  The concentration of albumin, wbc and uric acid in the subjects' blood samples
Lipid analysis | Baseline to 3 months
  The concentration of total cholesterol , triglyceride , HDL-cholesterol and LDL-cholesterol in the subjects' blood samples
Sugar test | Baseline to 3 months
  The concentration of fasting sugar and HbA1C in the subjects' blood samples
The quality of life | Baseline to 3 months
  It will measure by the Kidney Disease Quality of Life ([KDQOL]-SF™) questionnaire
Anemia test | Baseline to 3 months
  The concentration of hemoglobin (Hb) in the subject's blood samples
Urine protein analysis | Baseline to 3 months
  Urine specimen collection will be evaluated on the spot and 24-hour urine protein
24-hour Dietary recall | Baseline to 3 months
  There will be collected by food models or a photography atlas to estimate portion size
Gastrointestinal symptoms measures | Baseline to 3 months
  There will be collected by questionnaires symptoms or chief complaints
Grip strength levels | Baseline to 3 months
  Hand grip strength was measured by grip strength device
Blood gas | Baseline to 3 months
  The concentration of blood gas test in the subject's blood samples
Electrolytes Analysis | Baseline to 3 months
  The concentration of electrolytes analysis in the subject's blood samples
Mitochondrial oxidative stress | Baseline to 3 months
  The concentration analysis in the subject's blood or urine samples, such as MDA

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsu Chen, MDPHD, Principal Investigator — Division of Nephrology in Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, ROC, Taiwan